CLINICAL TRIAL: NCT03907917
Title: The Effects of Transcranial Direct Current Stimulation on Fear Extinction Learning and Memory Processes
Brief Title: Transcranial Direct Current Stimulation and Fear Extinction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Adams (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Thomas Adams, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1412015006_b; 1K23MH111977 (NIH)
Record Dates: First submitted 2019-04-01; First posted 2019-04-09 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to receive Active (real) or Sham (placebo) transcranial direct current stimulation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will be administrated by independent research staff. Double-blind software will be used to ensure that the experimenter and subject remain blind during task administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Current will be ramped in/out for 30 seconds at the begging and end of a 20-minute period and a constant current will be delivered for the 20-minutes between ramping.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): Current will be ramped in/out for 30 seconds at the begging and end of a 20-minute period during which no stimulation will be delivered.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Subjects will receive 20 minutes of multifocal transcranial direct current stimulation. The anode will be placed over the frontal pole (Fpz, 10-20 EEG) and will be surrounded by 5 return electrodes (cathodes). Current will be set at 1.5mA and will be ramped in/out at the begging and end of the 20-minutes of stimulation over the course of 30 seconds.
  Other Names: transcranial direct current stimulation; transcranial electrical stimulation; Starstim®

SUMMARY:
Psychiatric disorders characterized by pathological fear and anxiety are common and often disabling. Despite their limitations, exposure therapies are among the most efficacious treatments for these disorders. Extinction learning is thought to be a core mechanism of therapeutic exposure. Extinction learning is mediated by a well-defined circuit encompassing the medial prefrontal cortex (mPFC), amygdala, and hippocampus. This raises the exciting possibility that direct engagement of this circuitry might enhance the response to therapeutic exposure. Transcranial direct current stimulation (tDCS) is a neuromodulation technology that can augment brain plasticity, learning, and memory. The proposed study will evaluate whether tDCS can engage extinction circuitry, and improve extinction learning and memory.

This study will enroll psychiatrically healthy volunteers to test whether tDCS applied to the mPFC can augment spontaneous mPFC activity, engagement of extinction circuitry during extinction learning and recall, and classically-conditioned extinction learning and memory. Healthy volunteers will complete a standardized, three-day fear conditioning and extinction learning and memory task. On day 1, participants will complete a fear conditioning task. On day 2, participants will receive sham (placebo) or active tDCS prior to completing a fear extinction learning task. On day 3, participants will complete an extinction recall task. Electrodermal activity and heart rate will be continuously monitored during the conditioning and extinction procedures to assess autonomic arousal. All procedures will be completed in a magnetic resonance imaging (MRI) scanner; imaging data will be collected before and after tDCS and during all conditioning and extinction procedures.

DETAILED DESCRIPTION:
Most effective behavioral treatments of disordered anxiety involve repeated exposure to feared stimuli, which often results in systematic reductions in fearful responding to said stimuli. It is believed that this process results from successful fear extinction, a well-characterized learning process that is mediated by fear extinction brain circuitry. Namely, fear extinction is an inhibitory learning process that requires activation and plasticity within a variety of brain regions, including the medial prefrontal cortex (mPFC), which can exert inhibitory control over fearful responding and parts of the brain that drive said responding. Behavioral treatments of disordered anxiety, while effective, have serious limitations; many patients fail to respond at all or only partially respond to exposure-based treatments. One candidate reason for this is deficits in fear extinction learning or memory processes. The proposed study aims to examine the effects of non-invasive neuromodulation - namely, multifocal transcranial direct current stimulation (tDCS) targeting the mPFC - on spontaneous mPFC activity (Aim 1), functional activation of fear extinction circuitry (Aim 2), and fear extinction learning and memory (Aim 3).

This study will randomize 64 psychiatrically healthy volunteers at the Yale (proposed n = 32) and the University of Kentucky (proposed n = 32) for Aims 1-3. Following the completion of proper diagnostic and safety screening and Institutional Review Board (IRB) approved informed consent, healthy volunteers will complete a 3-day experimental procedure. Subjects will be conditioned to fear a previously neutral stimulus on Day 1. Subjects will be randomized (1:1, double-blind) to receive Active or Sham tDCS prior to fear extinction training on Day 2. Allocation will be done by independent research staff at Yale, who is experienced with such allocation, using block randomization (blocks of 8), stratified by sex. Subjects and investigators will be blind to allocation. Lastly, the strength of extinction recall will be tested on Day 3. Functional magnetic resonance imaging (fMRI) and psychophysiological measures (electrodermal activity and heart rate) will be acquired during all fear conditioning, extinction, and recall procedures and prior to and after tDCS.

tDCS will be delivered using an 8-channel Starstim transcranial electric stimulator from Neuroelectrics. To target the mPFC, the anodal electrode will be placed over the frontal pole (Fpz, 10-20 EEG landmarks) and will be surrounded by five return (cathodal) electrodes in a circumferential array (AF7, AF8, F3, Fz, and F4). Subjects in the Active tDCS condition will receive 20 minutes of direct current stimulation for 20 minutes; current will be ramped in and out for 30 seconds at the beginning and end of the 20-minute period. Subjects in the Sham tDCS condition will receive the same electrode placement and ramping procedures, but no current will be delivered between ramping.

All healthy volunteers will complete state-of-the-art Human Connectome Project Style (HCP-Style) accelerated multiband acquisition sequences. Scan sequences will be identical across sites. Scans will include a mixture of structural, resting state, and functional fMRI sequences. All scans will be completed on Siemens Prisma 3T scanners using 64-channel head coils. Psychophysiological measures will include electrodermal activity (EDA) and heart rate. All psychophysiological data will be collected with MRI-compatible Biopac systems.

Study 1 is well-powered for both planned and exploratory analyses; proposed methods help to improve signal-to-noise-ratio (SCR) and our proposed sample size of 64 will adequately power all a priori analyses, planned contrasts, and exploratory analyses. Power analysis suggested a sample of 42 would be adequate for the proposed primary hypothesis tests. We propose to recruit 70 participants to allow for approximately 10% attrition or data failures (e.g., head movement or null skin conductance response [SCR]). Our statistical approach and statistical power were developed in collaboration with statistical consultants of the PI and the primary mentor.

The proposed study will provide important preliminary data to examine the potential for medial prefrontal tDCS to augment and enhance fear extinction processes across multiple levels of analyses: the effects of tDCS on extinction circuitry and classically-conditioned extinction learning and memory.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent (as established by clinical interview), and voluntary, signed informed consent prior to the performance of any study-specific procedures;
* Ability and willingness to perform study-relevant clinical assessments;
* Ability and willingness to receive transcranial direct current stimulation (tDCS);
* Ability and willingness to complete magnetic resonance imaging (MRI) scans;
* Free of current psychiatric diagnosis;
* Psychiatrically healthy;
* 18-55 years of age;
* Medication free or stable (> 4 weeks) medication(s).

Exclusion Criteria:

* Any unstable medical, psychiatric, or neurological condition (including active or otherwise problematic suicidality) that may necessitate urgent treatment;
* Any substance dependence or severe substance abuse within the past 6 months;
* Daily use of psychotropic medications that substantially lower seizure threshold (e.g., clozapine);
* Daily use of psychotropic drugs that may interfere with extinction learning (e.g., anxiolytics);
* Any history of a psychotic disorder or of mania;
* Current active suicidal ideation or any suicidal intent;
* Any major neurological disease or history of major head trauma, including concussion with extended loss of consciousness, or of psychosurgery;
* Any history of epilepsy;
* Pregnancy;
* Any metal in the body or other contraindication to MRI scanning or tDCS;
* Any history of adverse effects to brain stimulation;
* A current Diagnostic and Statistical Manual diagnosis in the past 6 months, as determined by clinical interview;
* History of a severe psychiatric disorder, either documented or by clinician judgment;
* Use of drugs that are known to influence hemodynamic properties, except for drugs that are used to treat hypertension;
* Severe claustrophobia, back pain, or other condition that may make an extended magnetic resonance scan difficult or lead to excessive movement during the scan.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Fractional amplitude of low frequency fluctuations (fALFF) | Immediately following administration of tDCS on day 2 of the protocol.
  fALFF is a measure of resting brain activity that is derived by calculating regionally-specific fluctuations in Blood Oxygen Level-Dependent (BOLD) activation within a low-frequency band, typically while the participant is at rest.
Event related brain activation during extinction learning | BOLD imaging will be measured during extinction training on day 2 of the protocol.
  Blood Oxygen Level-Dependent imaging (BOLD imaging) will be measured during extinction training.
Event related brain activation during extinction recall | BOLD imaging will be measured during the test of extinction recall on day 3 of the experimental protocol.
  Blood Oxygen Level-Dependent imaging (BOLD imaging) will be measured during extinction recall.
Skin conductance response (SCR) during extinction learning | SCR will be measured during extinction learning on day 2 of the experimental protocol.
  SCR will be measured by collecting electrodermal activity (EDA) on the left hand and subtracting the maximal EDA value during the presentation of the virtual context (CX) picture from the maximal EDA value during the presentation of the conditioning stimuli (CS).
Skin conductance response (SCR) during extinction recall | SCR will be measured during extinction recall on day 3 of the experimental protocol.
  SCR will be measured by collecting electrodermal activity (EDA) on the left hand and subtracting the maximal EDA value during the presentation of the virtual context (CX) picture from the maximal EDA value during the presentation of the conditioning stimuli (CS).

SECONDARY OUTCOMES:
Functional connectivity measure of tDCS | Immediately prior to and following administration of tDCS. Change in connectivity from pre to post stimulation (delta) will be modeled and used as the dependent variable.
  Correlations between brain regions over the time course.
Functional connectivity during extinction learning | During extinction learning on day 2 of the experimental protocol.
  Correlations between brain regions over the time course
Functional connectivity during extinction recall | During extinction recall on day 3 of the experimental protocol.
  Correlations between brain regions over the time course

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Adams, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - Yale School of Medicine, New Haven, Connecticut
  - University of Kentucky, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
Raw imaging and psychophysiological data will be freely available upon study publication. Data will be stored on a yet to be determined data sharing repository supported by the National Institutes of Health.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available following study publication.

DOCUMENTS (1):
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT03907917/ICF_000.pdf